CLINICAL TRIAL: NCT05882227
Title: Nursing Intervention for the Reduction of Anxiety During the Process of Primary Total Hip Arthroplasty Within the Optimized Recovery Program.
Acronym: NIRARATC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Elisabet Ripoll, Principal investigator, University of Barcelona
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2023/0015; Jordi Galimany Masclans (Other: Barcelona University); Zaida Palmira Agüera Imbernón (Other: Barcelona University); Montserrat Puig Llobet (Other: Barcelona University)
Record Dates: First submitted 2023-04-23; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthrosis; ERAS; Anxiety; Nurse
Keywords: hip arthroplasty; ERAS; Nursing care
MeSH Terms: conditions — Osteoarthritis; Anxiety Disorders | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): patients will watch a video with discharge information taken from the document "Optimized hip replacement recovery program; information for patients, family members or caregivers".
  Interventions: Behavioral: video
- Traditional information (Active Comparator): patients will receive discharge information will be provided through the document entitled "Optimized Hip Replacement Recovery Program; Information for Patients, Family or Caregivers".
  Interventions: Behavioral: Traditional information

INTERVENTIONS:
Behavioral: video — The patients will receive the discharge information through the visualization of a video with discharge information extracted from the optimized hip prosthesis recovery program document; information for patients, relatives or caregivers. The video will consist of two parts: a first part where it will be explained what will happen in the next hours in the unit, the documentation that will be delivered at discharge and the pharmacological treatment. The second part will consist of a video explaining wound care at discharge, discharge recommendations, symptoms that may appear after surgery and alarm symptoms.
  Arms: Video
Behavioral: Traditional information — Patients will receive the information at discharge by means of the document entitled "Optimized Hip Replacement Recovery Program; information for patients, relatives or caregivers", which will act as a control group.
  Arms: Traditional information

SUMMARY:
Osteoarthrosis (OA) is a chronic, degenerative disease characterized by joint wear and tear. It is a major cause of pain, disability and decreased quality of life. Total hip arthroplasty (THA) and total knee arthroplasty (TKA) represent an effective alternative for the treatment and pain control of patients with osteoarthritis. The "fast-track" program is translated as enhanced recovery or fast-track, and consists of the active participation of patients in their own recovery and immediate post-surgical mobilization, thanks to preoperative education through an educational workshop, the type of analgesia used and the empowerment of the patient in his or her own recovery.

The problem of anxiety in the surgical patient and the role of nurses in it has been widely studied for some decades, as shown in the scientific literature. Our experience as professionals of a hospital unit of orthopedic surgery and traumatology shows us the reality of this situation and the investigators find that when discharging patients who have undergone surgery and are discharged after 24 hours, the patient almost globally manifests a series of expressions, behaviors or behaviors that are related to anxious behavior, a completely natural human response of a patient who does not know what he is going to face. This leads us to detect a need to reinforce the information provided at discharge and the accompaniment during the first weeks after discharge.

Anxiety is a complex reaction to potentially dangerous situations or stimuli. It is an alarm signal that triggers a series of responses to cope with the situation. Anxiety is an emotional response that encompasses unpleasant cognitive aspects and physiological alterations that manifest themselves with high nervousness and even motor alterations.

Surgery is perceived by the patient as an important stress factor that can translate into nervousness and anxiety. Anxiety is almost always present during surgery, to a greater or lesser degree, both preoperatively and postoperatively.

Several studies have shown that good preoperative information reduces preoperative and postoperative anxiety. Patients need information about their process since dispelling their doubts will minimize anxiety. Currently there is very little information on anxiety during the whole surgical process. Therefore, in the present project the investigators propose to carry out a research study to analyze whether nursing intervention has beneficial results in the surgical patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled with signed consent for primary hip arthroplasty surgery, age over 18 years, patients who agree to participate in the study.

Exclusion Criteria:

* Patients who are discharged to a social-health center, patients with cognitive or mental disorders, patients who cannot read or write.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Before the surgical intervention during the visit with the advanced practice nurse (APN) who will measure the pre-intervention outcome.
  HADS is a self-report questionnaire designed to screen anxious and depressive states in patients in non-psychiatric settings. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately.
Hospital Anxiety and Depression Scale (HADS) | 24 hours after surgery just prior to discharge from the hospital.
  HADS is a self-report questionnaire designed to screen anxious and depressive states in patients in non-psychiatric settings. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately.
Hospital Anxiety and Depression Scale (HADS) | One month after surgery when patiente comes to visit the doctor.
  HADS is a self-report questionnaire designed to screen anxious and depressive states in patients in non-psychiatric settings. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately.
Hospital Anxiety and Depression Scale (HADS) | six months after surgery when patiente comes to visit the doctor.
  HADS is a self-report questionnaire designed to screen anxious and depressive states in patients in non-psychiatric settings. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately.
Hospital Anxiety and Depression Scale (HADS) | A year after surgery just prior to discharge from the hospital.
  HADS is a self-report questionnaire designed to screen anxious and depressive states in patients in non-psychiatric settings. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately.
EuroQol-5D | Before the surgical intervention during the visit with the advanced practice nurse (APN) who will measure the pre-intervention outcome.
  The EQ-5D family of instruments have been developed to describe and value health across a wide range of disease areas. They are also frequently used in research into health in the general population. The EQ-5D-3L essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale.The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
EuroQol-5D | 24 hours after surgery just prior to discharge from the hospital.
  The EQ-5D family of instruments have been developed to describe and value health across a wide range of disease areas. They are also frequently used in research into health in the general population. The EQ-5D-3L essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale.The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
EuroQol-5D | One month after surgery when patiente comes to visit the doctor.
  The EQ-5D family of instruments have been developed to describe and value health across a wide range of disease areas. They are also frequently used in research into health in the general population. The EQ-5D-3L essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale.The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
EuroQol-5D | six months after surgery when patiente comes to visit the doctor.
  The EQ-5D family of instruments have been developed to describe and value health across a wide range of disease areas. They are also frequently used in research into health in the general population. The EQ-5D-3L essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale.The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
EuroQol-5D | a year after surgery when patiente comes to visit the doctor.
  The EQ-5D family of instruments have been developed to describe and value health across a wide range of disease areas. They are also frequently used in research into health in the general population. The EQ-5D-3L essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale.The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.

SECONDARY OUTCOMES:
Sociodemographic variables | These variables will be collected 24 hours after surgery just prior to discharge from the hospital.
  Sex and age.

CONTACTS AND LOCATIONS:
Overall Officials: Zaida Agüera, Nurse, Study Director — barcelona University
Locations (1):
- Elisabet Ripoll Romero, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montin L, Suominen T, LeiniKilpi H. The experiences of patients undergoing total hip replacement. Journal of Orthopaedic Nursing. 2002 febrer; 6(1): 23-29.
- [Background] Montin L, Suominen T, Leino-Kilpi H.The experiences of patients undergoing total hip replacement. Journal of Orthopaedic Nursing.2002;6(1):23-29.
- [Background] his document should be cited as: EuroQol Research Foundation. EQ-5D-3L User Guide, 2018. Available from: https://euroqol.org/publications/user-guides.
- [Background] Stern AF. The hospital anxiety and depression scale. Occup Med (Lond). 2014 Jul;64(5):393-4. doi: 10.1093/occmed/kqu024. No abstract available. PMID 25005549